CLINICAL TRIAL: NCT03549715
Title: NEoadjuvant Dose-dense MVAC In cOmbination With Durvalumab (MEDI4736) and Tremelimumab in Muscle-invasive Urothelial Carcinoma
Brief Title: NEoadjuvant Dose-dense MVAC In cOmbination With Durvalumab and Tremelimumab in Muscle-invasive Urothelial Carcinoma
Acronym: NEMIO
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Association Pour La Recherche des Thérapeutiques Innovantes en Cancérologie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEMIO
Record Dates: First submitted 2018-05-15; First posted 2018-06-08 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Infiltrating Bladder Urothelial Carcinoma
MeSH Terms: interventions — durvalumab; tremelimumab; M-VAC protocol

STUDY DESIGN:
Intervention Model Description: The sample size will be balanced between 2 arms. Initially, 12 patients (6 in each arm) will be included and randomized between durvalumab + ddMVAC (ARM A) or durvalumab + tremelimumab + ddMVAC (ARM B)
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A: durvalumab + ddMVAC (Experimental): Durvalumab + ddMVAC Durvalumab 1500 mg IV D1 every 28 days Durvalumab will be administered at the hospital every 28 days prior to administration of ddMVAC on D1.
  Interventions: Drug: Durvalumab; Drug: MVAC Protocol
- ARM B: durvalumab + tremelimumab+ ddMVAC (Experimental): durvalumab + tremelimumab + ddMVAC Tremelimumab 75 mg IV D1 every 28 days Tremelimumab will be administered first, with durvalumab infusion starting approximately 1 hour (maximum 2 hours) after the end of the tremelimumab infusion.
  Infusion of ddMVAC will start approximately 1 hour after completion of durvalumab.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: MVAC Protocol

INTERVENTIONS:
Drug: Durvalumab — 1500 mg IV D1 every 28 days (2 doses for each patient)
  Other Names: MEDI4736
Drug: Tremelimumab — 75 mg IV D1 every 28 days ((2 doses for each patient)
  Other Names: CP-675,206
  Arms: ARM B: durvalumab + tremelimumab+ ddMVAC
Drug: MVAC Protocol — 1. Methotrexate 30 mg/m2 IV D1
  2. Vinblastine 3 mg/m2 IV D1
  3. Adriamycin (doxorubicin) 30 mg/m2 IV D1
  4. Cisplatin 70 mg/m2 IV D1
  Other Names: ddMVAC

SUMMARY:
This is an open label, phase I/II clinical trial to evaluate the efficacy and safety of 2 cycles of durvalumab without (Arm A) or with (Arm B) tremelimumab in association with ddMVAC as neoadjuvant therapy in patients with MIUC.

DETAILED DESCRIPTION:
Study Population:

Patients with MIUC fit to receive cisplatin.

Study Design:

The trial is designed as a non-comparative, open-label phase I/II study.

Divided in two phases:

The run In phase (I) and a phase II study. During the run-in phase, a limited number of patients (n=12-18) will be treated with durvalumab + ddMVAC or durvalumab + tremelimumab + ddMVAC (6-9 patients each). If the toxicity rate is acceptable (not higher than 2 out of 6 or 3 out of 9 patients per arm) the study will continue as a randomized phase II study. During phase II, the efficacy and safety of durvalumab + ddMVAC and durvalumab + tremelimumab + ddMVAC

Research hypothesis:

Combination of checkpoint inhibitors (CPI), durvalumab ± tremelimumab, with neoadjuvant ddMVAC will improve the pathological complete response (pCR) rate in patients with muscle-invasive urothelial carcinoma (MIUC). No additional toxicity of the combination CPI + ddMVAC is expected.

Investigational Product(s):

Durvalumab: 1500 mg IV D1 every 28 days Durvalumab will be administered at the hospital every 28 days prior to administration of ddMVAC on D1.

Tremelimumab 75 mg IV D1 every 28 days Tremelimumab will be administered first, with durvalumab infusion starting approximately 1 hour (maximum 2 hours) after the end of the tremelimumab infusion.

Translational research:

Mechanism of response/resistance to neoadjuvant treatment will be assessed by comparing molecular and immunological tumor profiles before treatment (transurethral resection tumor samples) and after treatment (cystectomy samples). In addition, circulating tumor DNA (ctDNA) and urine tumor DNA (utDNA) will be analysed during treatment (ctDNA and utDNA) and after surgery (ctDNA).

Immunological profiles will be established using a specific metagene signature for major cell types of the tumor microenvironment and chemokines, cytokines and regulatory molecules , and will be validated using relevant markers by immunohistochemistry (IHC) on formalin-fixed paraffin-embedded (FFPE) tumor sections.

Metabolomic profiling will also be conducted by analyzing metabolites present in urinary samples with a Proton-based nuclear magnetic resonance (1H-NMR), and correlations with prognosis, molecular profile or/and with immunological signature determined.

Finally, correlations between tumor pathological factors (e.g., pTNM, nuclear grade, variant squamous differentiation or sarcomatoid dedifferentiation) and prognosis will be evaluated using IHC on FFPE tissue sections.

Sample Size: Approximately 121 patients are planned to be included.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally required authorization (e.g., EU Data Privacy Directive in the EU) obtained from the patient prior to performing any protocol-related procedures, including screening evaluations
2. Age ≥18 years at time of study entry
3. Histologically confirmed MIUC (also termed TCC) of the bladder. Patients with mixed histologies are required to have a dominant transitional cell pattern (urothelial carcinoma must be > 50%)
4. Localized MIUC of the bladder with clinical stage T2-T4a and ≤N1 disease ( the single lymph node must be < 15 mm (short axis) on imaging
5. Patients with urothelial carcinoma of the prostatic urethra
6. Bodyweight >45kg
7. Patients eligible for cisplatin-based neoadjuvant chemotherapy, including:

   * Creatinine clearance (CL) >60 mL/min based on the Modification of Diet in Renal Disease Study (MDRD) formula
   * Cardiac left ventricular ejection fraction (LVEF) ≥50%
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
9. Absence of metastasis, as confirmed by a negative baseline CT or MRI scan of the pelvis, abdomen, and chest no more than 4 weeks prior to randomization. Patients with clinical stage N1 disease are eligible if the single lymph node measures ≤2 cm in greatest dimension.
10. Adequate organ and marrow function as defined below (obtained within 14 days prior to the first study treatment):

    * Hemoglobin ≥10.0 g/dL (patients may be transfused to meet this criterion)
    * Absolute neutrophil count (ANC) ≥1500 cells/μL (without G-CSF support within 2 weeks prior to Cycle 1, Day 1)
    * WBC counts >2500/µL
    * Platelet count ≥100,000/µL (without transfusion within 2 weeks prior to Cycle 1, Day 1)
    * Serum bilirubin ≤1.0 x institutional upper limit of normal (ULN). Patients with known Gilbert disease who have serum bilirubin level ≤3 x ULN may be enrolled.
    * AST, ALT, and alkaline dehydrogenase ≤2.5 x ULN
    * Partial thromboplastin time/prothrombin time (PTT/PT) ≤1.5 x ULN or international normalized ratio (INR) <1.7 x ULN
11. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
    * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
12. Women of childbearing potential and non-sterilized males who are sexually active with a female partner of childbearing potential must be willing to use contraceptive methods during the treatment period and for at least 6 months after the last dose of treatment
13. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Urothelial carcinoma of the upper tract
2. Any approved anti-cancer therapy for urothelial carcinoma, including chemotherapy, or immunotherapy prior to initiation of study treatment. Of note, previous intravesical BCG injections are allowed if administered for non-muscle invasive urothelial carcinoma
3. Primary chemoradiation for bladder preservation for urothelial carcinoma of the bladder
4. Impaired renal function (glomerular filtration rate [GFR]<60 mL/min); GFR should be assessed by calculation from serum/plasma creatinine (MDRD formula)
5. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
6. Grade 2 or greater hearing loss that contraindicates cisplatin use. Threshold shift of >25 decibel averaged at 2 contiguous test frequencies in least one ear.

   Exception: Patients with Grade 2 hearing loss diagnosed on the audiogram that are asymptomatic (no complain of hearing loss and no tinnitus) can be enrolled in the study.
7. Grade 2 or greater peripheral neuropathy
8. Oral anticoagulation treatment (vitamin K antagonist should be replaced by low-molecular-weight heparin).
9. Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days or five half-lives of the drug
10. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
11. Any concurrent chemotherapy, investigational product, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable
12. Major surgical procedure (as defined by the Investigator) other than for diagnosis within 28 days prior to Cycle 1
13. History of prior organ transplantation, including stem cell allografting
14. History of autoimmune disease, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone and type I diabetes mellitus on stable dose of insulin may be eligible for this study
15. All micropapillary and plasmacytic forms, with or without squamous cell adenocarcinoma
16. Severe infections within 4 weeks prior to Cycle 1, Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
17. Signs or symptoms of infection within 2 weeks prior to Cycle 1, Day 1
18. Receipt of therapeutic oral or IV antibiotics within 2 weeks prior to Cycle 1, Day 1
19. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within the previous 6 months, unstable arrhythmias, or unstable angina
20. History of another primary malignancy within 3 years prior to Cycle 1, Day 1, except for:

    Localized low-risk prostate cancer (defined as Stage ≤T2b, Gleason score ≤7, and prostate-specific antigen [PSA] at prostate cancer diagnosis ≤20 ng/mL [if measured]) treated with curative intent and without PSA recurrence Low-risk prostate cancer (defined as Stage T1/T2a, Gleason score <7, and PSA ≤10 ng/mL) who are treatment-naive and undergoing active surveillance Patients with malignancies of a risk of metastasis/death (e.g., risk of metastasis or death <5% at 5 years) are eligible after investigator's approval if they meet both of the following criteria: Malignancy treated with expected curative intent, and no evidence of recurrence or metastasis by follow-up imaging and any disease-specific tumor markers
21. History of leptomeningeal carcinomatosis
22. History of idiopathic pulmonary fibrosis, organizing pneumonia
23. Serum albumin <25 g/L
24. LVEF <50%
25. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 electrocardiograms (ECGs) within 15 minutes at 5 minutes apart
26. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if PCR is negative for HCV RNA
27. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

    Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection) Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
28. Receipt of live attenuated vaccine within 30 days prior to the first dose of study treatment. Note: Patients, if enrolled, should not receive live vaccine whilst receiving study treatment and for up to 30 days after the last dose of study treatment
29. Female patients who are pregnant or breastfeeding, or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab + tremelimumab combination therapy
30. Known allergy or hypersensitivity to chimeric or humanized antibodies or fusion proteins, or to any of the study drugs or study drug excipients
31. Prior randomisation or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment
32. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that, in the opinion of the Investigator, makes the patient unsuitable for participation in the study Procedures for withdrawal of incorrectly enrolled patients are presented in Section 4.3 If a patient withdraws from participation in the study, then his or her enrollment/randomization code cannot be reused. Withdrawn patients will not be replaced.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Toxicity Grade | 68 months
  Grade ≥ 3 treatment related toxicity rate
pathologic complete response | 1 year
  pCR rate after ddMVAC + durvalumab ± tremelimumab period

SECONDARY OUTCOMES:
Disease-Free Survival (DFS) | 2 years
  To evaluate the 2-year disease-free survival (DFS) rate.
Overall Survival (OS) | 2 years
  To evaluate the 2-year overall survival (OS) rate
Adverse Events (AEs). | 68 months
  To evaluate the incidence of adverse events (AEs).
Pathologic downstaging | During procedure
  To evaluate the pathologic downstaging rate (defined as the presence of residual tumor ≤T1 on cystectomy, excluding T0).

OTHER OUTCOMES:
Molecular profile | 2 years
  To determine changes in the molecular profile and immunological signature of the tumor after treatment compared with before treatment.
Factors of pCR | 1 year
  To identify predictive factors of pCR response to treatment.
Immunological signature | 2 years
  To determine changes in the immunological signature of the tumor after treatment compared with before treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Constance THIBAULT, MD, Principal Investigator — Hôpital Européen Georges Pompidou, Oncology department of Pr Stéphane OUDARD
Locations (15):
- France (15):
  - Hôpital Saint André, CHU de Bordeaux, Bordeaux
  - Sasu Roc37, Chambray-lès-Tours
  - CHU Henri-Mondor, Créteil
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Antoine Lacassagne, Nice
  - Groupe Hospitalier Pitié-Salpetrière, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Cochin, Paris
  - Centre Eugène Marquis, Rennes
  - Hia Begin, Saint-Mandé
  - Hôpitaux universitaires de Strasbourg, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
  - Hôpital Européen Georges Pompidou, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No
No plan to share

REFERENCES:
- [Derived] Thibault C, Elaidi R, Vano YA, Rouabah M, Braychenko E, Helali I, Audenet F, Oudard S. Open-label phase II to evaluate the efficacy of NEoadjuvant dose-dense MVAC In cOmbination with durvalumab and tremelimumab in muscle-invasive urothelial carcinoma: NEMIO. Bull Cancer. 2020 Jun;107(5S):eS8-eS15. doi: 10.1016/S0007-4551(20)30281-2. PMID 32620213